CLINICAL TRIAL: NCT06425601
Title: The Impact of Chest Drain Type on Pain, Drainage Efficacy and Short Term Outcome Following VATS Lobectomy for Lung Cancer: A Prospective Randomized Study Comparing Silicone Versus PVC Drains
Brief Title: A Comparison of Silicone Versus Polyvinylchloride (PVC) Drains Following VATS Lobectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Boris Greif, MD, Head of Thoracic Surgery, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0120-445/2019/8
Record Dates: First submitted 2024-05-08; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Postoperative Pain; Postoperative Complications
Keywords: VATS; lung lobectomy; postoperative pain; chest drain; analgesia
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications; Agnosia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silicone (SIL) group (Experimental): For postoperative pleural space drainage a silicone coaxial drain of size French 24 (Redax Coaxial Drain, Redax S.p.A., Poggio Rusco Mantova, Italy) was used
  Interventions: Device: SIL drain
- PVC group (Active Comparator): For postoperative pleural space drainage a standard polyvinyl chloride drain of size French 24 (Argyle, Covidien, Mansfield, USA) was used
  Interventions: Device: PVC drain

INTERVENTIONS:
Device: SIL drain — Silicone chest tube used for pleural space drainage after VATS lobectomy
  Arms: Silicone (SIL) group
Device: PVC drain — Polyvinyl chloride chest tube used for pleural space drainage after VATS lobectomy
  Arms: PVC group

SUMMARY:
The goal of this prospective randomized clinical trial is to compare the impact of the chest tube type on pain, chest drainage efficacy and early postoperative outcome following VATS lobectomy for lung cancer.

The main questions it aims to answer are:

* silicone chest drains are less painful compared to standard PVC drains?
* is there any difference in chest drainage efficacy and short term outcome between the two groups? Researchers will compare silicone chest drain group with PVC chest drain group to see if there is any difference in postoperative pain, chest drainage efficacy and short term outcome.

ELIGIBILITY:
Inclusion Criteria:

* primary lung cancer eligible for VATS lobectomy by tumor board meeting

Exclusion Criteria:

* age under 18 years
* high risk of post-operative complications (ASA > 3, diffusion capacity for transfer factor (TLCO) or forced expiratory volume at one second (FEV1) ≤ 40%, cycle ergometry with oxygen consumption (VO2 max) < 15 ml/kg/min)
* tumors growing in parietal pleura
* extended lung resection diffuse
* previous surgery in the same hemithorax
* chronic pain
* chronic use of analgesics or sedatives
* surgical revision
* inability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Analgesics consumption | 2 days
  Amount of analgesics used first two days after the surgery was analyzed and reported in milligrams. Higher scores mean a worse outcome.
Need for peroral analgesia after the chest tube removal | 2 days
  Need for peroral analgesia at first, second and fourth week after chest tube removal was assessed and reported as frequency in number. Higher scores mean a worse outcome.
Maximal inspiratory pressure | 2 days
  Post-operative pain during the first two days after the surgery was analyzed by measuring the maximal inspiratory pressure (MIP) in cmH2O. Higher scores mean a better outcome.
Maximal expiratory pressure | 2 days
  Post-operative pain during the first two days after the surgery was analyzed by measuring the maximal expiratory pressure (MEP) in cmH2O. Higher scores mean a better outcome.
Visual analogue scale | 2 days
  Post-operative pain during the first two days after the surgery was analyzed by using the visual analogue scale (VAS). Scale tittle was Visual Analogue Scale. Minimum value on a scale was 0 and maximum value was 10. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Duration of chest drainage | 1 month
  The effectiveness of chest drainage was analyzed by assessing the duration of chest drainage in days. Higher scores mean a worse outcome.
Pneumothorax rate on the day of surgery | First day
  The effectiveness of chest drainage was analyzed by assessing the rate of pneumothorax (frequency in number) on chest x-ray on the day of surgery. Higher scores mean a worse outcome.
Pneumothorax rate after chest tube removal | 1 month
  The effectiveness of chest drainage was analyzed by assessing the rate of pneumothorax (frequency in number) on chest x-ray after removal of the drain. Higher scores mean a worse outcome.
Pleural effusion rate on the day of surgery | First day
  The effectiveness of chest drainage was analyzed by assessing the rate of pleural effusion (frequency in number) on chest x-ray on the day of surgery. Higher scores mean a worse outcome.
Pleural effusion rate after chest tube removal | 1 month
  The effectiveness of chest drainage was analyzed by assessing the rate of pleural effusion (frequency in number) on chest x-ray after removal of the drain. Higher scores mean a worse outcome.
Subcutaneous emphysema rate | 1 month
  The effectiveness of chest drainage was analyzed by assessing the rate of clinically expressed subcutaneous emphysema (frequency in number). Higher scores mean a worse outcome.
Prolonged air leak rate | 1 month
  The effectiveness of chest drainage was analyzed by assessing the rate of prolonged air leak over 5 days (frequency in number). Higher scores mean a worse outcome.
Reintervention rate | 1 month
  The effectiveness of chest drainage was analyzed by assessing the rate of reintervention (thoracentesis or chest drainage) after chest tube removal (frequency in number). Higher scores mean a worse outcome.
Duration of hospital stay | 1 month
  Early postoperative course was analyzed by assessing the duration of hospital stay (in days). Higher scores mean a worse outcome.
Respiratory complication rate | 1 month
  Early postoperative course was analyzed by assessing the rate of respiratory complications (frequency in number). Higher scores mean a worse outcome.
Readmission rate | 1 month
  Early postoperative course was analyzed by assessing the rate of readmission in the first month after drain removal (frequency in number). Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Boris Greif, Principal Investigator — UMC Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Derived] Greif B, Zgajnar J, Stupnik T. Impact of chest tube type on pain, drainage efficacy, and short-term treatment outcome following video-assisted thoracoscopic surgery lobectomy: a randomized controlled trial comparing coaxial silicone drains and standard polyvinyl chloride drains. J Thorac Dis. 2025 Feb 28;17(2):932-943. doi: 10.21037/jtd-24-1489. Epub 2025 Feb 21. PMID 40083488